CLINICAL TRIAL: NCT01018316
Title: UMOX - New Device for Oropharyngeal Preoxygenation
Status: Completed | Type: Observational
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Louis-Philippe Fortier, MSc, MD,FRCPC, Maisonneuve-Rosemont Hospital affiliated to the University of Montreal
Other Study IDs: HMR-MEM
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: Preoxygenation
Keywords: preoxygenation; UMOX

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The UMOX is a device that has been designed as an alternative to the conventional face mask for preoxygenation to be used when an optimal preoxygenation with a facemask is difficult to achieve(i.e: when a leak is present. A previous study in our hospital (unpublished data) has shown that the UMOX was only as effective as the conventional mask when a nose clip was used to prevent the patients from breathing in some air through the nose, thus preventing the dilution/contamination of the 100% oxygen delivered.In that study, the verbal indication giving to the subjects to breathe through the mouth was better than no indication at all but still yielded unsatisfactory results.

For this reason, the present study was designed to verify the hypothesis that while using the UMOX for preoxygenation, the verbal indication of breathing 8 vital capacity breaths added to the indication of breathing through the mouth would bring equivalent results -measured by the expired fraction of oxygen- as a preoxygenation of normal tidal breathing through a facemask during 3 to 5 minutes.

Preoxygenation was performed with the 60 volunteers placed in the supine position with 100% oxygen. All volunteers went though preoxygenation with two techniques: 1) breathing normal tidal volumes at a normal respiratory rate for a period of 5 minutes through a tight fitting conventional face mask, and 2) eight deep breaths (i.e. vital capacity breaths) through the UMOX device with verbal indication to use only the mouth to breathe.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II, smoker or non smoker

Exclusion Criteria:

* patients under 18 years old or over 65 years old; edentulous patients or those with craniofacial malformations, beards or mustaches; patients that have >30 kg over their ideal weight; and patients with moderate to severe pulmonary pathology

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada